CLINICAL TRIAL: NCT03964428
Title: Decreased Ferritin And Increased Hepcidin Serum Levels In Periodontitis Patients With Diabetes Mellitus Type 2. Controlled Before-And-After Study
Brief Title: Serum Ferritin and Hepicidin Concentration in Chronic Periodontitis Patients With T2DM
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Nayroz Abdel Fattah Mohamed Tarrad, lecturer, Fayoum University
Other Study IDs: fayoum dentistry
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Periodontitis; Type2 Diabetes
Keywords: periodontitis; ferritin; hepicidin; type 2 diabetes mellitus; non surgical perioontal therapy
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- periodontitis
- periodontitis with T2DM
- control

SUMMARY:
serum level of ferritin and hepicidin were evaluated in periodontitis patient with and without type 2 diabetes before and after non surgical periodontal treatment to clarify their in periodontal disease

ELIGIBILITY:
Inclusion Criteria:

* patients with more than 30% of the sites had clinical attachment level (CAL) 3-4mm with T2DM
* systemically healthy patients with more than 30% of the sites had clinical attachment level (CAL) 3-4mm
* healthy subjects had clinically healthy gingiva with ≤ 3mm pocket probing depth (PPD), nearly zero plaque index (PI), gingival index (GI), zero CAL.

Exclusion Criteria:

* (I) Pregnancy or lactation, (II) History of receiving professional periodontal treatment during the past 6 months; (III) Treatment with any type of medications and/ or antibiotics during the past 3 months and (IV) Current or former smokers.

Ages: 30 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: participants were collected from the Outpatient Clinic, Department of Oral Medicine, Periodontology and Diagnosis, and the restorative clinic for the control subjects, Faculty of Oral and Dental Medicine, fayoum University
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
ferritin concentration | 0-3 months
  ng/ml
hepicidin concentration | 0-3 months
  ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Nayroz Abelfattah Tarrad, Cairo, Egypt